CLINICAL TRIAL: NCT02909504
Title: Biomarkers in Mononuclear Blood Cells for Lithium Treatment Response of Bipolar Disorder
Brief Title: Gao NARASD Lithium Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Keming Gao (Other)
Collaborators: CellPrint Biotechnology (Other); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor-Investigator, Keming Gao, Clinical Director, Mood Disorders Program, UH Cleveland Medical Center, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-16-05
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium (Other): Eligible patients will receive lithium 300 mg twice daily and titrated in 300 mg increments every 7 days as tolerated to levels > 0.6 mEq/L
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — Eligible patients will receive lithium 300 mg twice daily and titrated in 300 mg increments every 7 days as tolerated to levels > 0.6 mEq/L

SUMMARY:
This study is a 4-month open-label study of lithium in the acute treatment of patients with bipolar I or II disorder. Eligible patients will receive lithium 300 mg twice daily and titrated in 300 mg increments every 7 days as tolerated to levels > 0.6 mEq/L. Blood samples are collected at baseline and at the end of study. Analyses of 45 molecule expressions in mononuclear blood cells at baseline and endpoint will be carried out after the completion of study. Fifty patients meeting Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria for bipolar I or II will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, subjects must meet all of the following criteria:

1. Able to provide informed consent before beginning any study-specific procedures;
2. Male or female, 18-70 years old;
3. Meets current DSM-5 criteria for bipolar I or II disorder as assessed by the The M.I.N.I. International Neuropsychiatric Interview (MINI);
4. Any symptomatic phase of bipolar I or II disorder including, depressive, manic, mixed or hypomanic
5. Global Clinical Impression-Severity for Bipolar Disorder (CGI-S-BD) ≥3;
6. Willing to take lithium;
7. If a sexually active female of childbearing potential, be using a reliable method of contraception;
8. Women with reproductive potential must have a negative urine pregnancy test;
9. Willing to have blood drawn:

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Unwilling to comply with study requirements;
2. Renal impairment (serum creatinine >1.5 mg/dL);
3. Thyroid stimulating hormone (TSH) over >20% above the upper normal limit (participants maintained on thyroid medication must be euthyroid for at least 3 months before Visit 1;
4. Other contraindication to lithium,
5. Patients who have had severe adverse reaction to Lithium;
6. Patients who require inpatient care;
7. Drug/alcohol dependence requiring immediate acute detoxification;
8. Pregnancy as determined by serum pregnancy test or breastfeeding;
9. History of nonresponse to lithium at doses ≥ 900 mg/d for ≥ 8 weeks;
10. Unwilling to have blood drawn
11. Patients with chronic medical conditions such as diabetes, coronary artery disease, immune diseases, infectious diseases and neurological disorders;
12. Active suicidal ideation with a plan or intent, a suicide attempt within past 6 months or more than 2 suicide attempts within the past 2 years.
13. Currently on lithium

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keming Gao, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center Department of Psychiatry, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lithium
Started | 24
Completed | 12
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 4
Not completed — Pregnancy | 1
Not completed — Subject moved | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lithium
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24
Bipolar Diagnosis [Count of Participants; unit: Participants]
  Bipolar I Disorder | 17
  Bipolar II Disorder | 7
Lifetime Generalized Anxiety Disorder (GAD) Diagnosis [Count of Participants; unit: Participants] | 16
Lifetime Social Phobia Diagnosis [Count of Participants; unit: Participants] | 13
Lifetime Attention Deficit Hyperactivity Disorder (ADHD) Diagnosis [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Expression of ~45 Molecules in Blood Cells of Patients With Bipolar I or II Disorder Being Treated With Lithium
Description: Molecule expression is measured as a function of relative fluorescence intensity. The number derives from a photomultiplier tube which essentially counts photons. Higher numbers mean a higher intensity. The values in the results tables represents change in fluorescence intensity between Baseline and Week 16 across various molecules of interest and compares responders (those who experience a >=50% decrease in mood symptom severity between baseline and week 16) and non responders (those who did NOT experience a >=50% decrease in mood symptom severity between baseline and week 16). The rows represent the various molecules that were analyzed.
Time Frame: Baseline and Week 16
Population: While we planned to analyze ~45 molecules of interest, poor quality of antibodies to some proteins & financial limitations limited us to only 28 proteins. The number of participants analyzed for protein expression differs from baseline characteristic and varies below as not all subjects had high enough levels of a particular protein to be analyzed.
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Groups:
- Lithium Non Responders; Lithium Responders: Lithium: Eligible patients will receive lithium 300 mg twice daily and titrated in 300 mg increments every 7 days as tolerated to levels > 0.6 mEq/L.
Arm/Group | Lithium Non Responders | Lithium Responders
Number analyzed (Participants) | 9 | 12
fluorescence intensity
  NLRP3 | 30.73 (5.66) | 26.00 (7.25)
  PDEB4: number analyzed (Participants) | 4 | 10
  PDEB4 | 28.15 (9.12) | 27.31 (5.78)
  BAK | 11.16 (2.08) | 11.50 (2.88)
  p-Fyn Yes | 12.49 (4.46) | 13.33 (6.44)
  HMGB1: number analyzed (Participants) | 6 | 11
  HMGB1 | 23.18 (8.69) | 22.61 (6.58)
  IRS2 | 25.29 (5.64) | 24.06 (8.71)
  p-CREB | 30.78 (4.34) | 30.46 (6.55)
  PPAR g | 21.90 (4.31) | 21.13 (5.62)
  TNFAIP3 | 33.74 (6.16) | 31.17 (6.64)
  TPH1 | 7.13 (1.04) | 7.23 (2.47)
  PKC theta: number analyzed (Participants) | 4 | 9
  PKC theta | 33.8 (7.11) | 35.81 (8.71)
  Bcl-2: number analyzed (Participants) | 9 | 11
  Bcl-2 | 39.72 (6.89) | 35.87 (8.94)
  iNOS | 24.51 (4.38) | 24.54 (7.54)
  NR3C1: number analyzed (Participants) | 4 | 8
  NR3C1 | 7.33 (2.16) | 6.69 (2.64)
  mTor | 22.87 (6.41) | 21.07 (8.60)
  PKA C-a | 24.51 (5.69) | 23.93 (7.08)
  Bcl-2 A1 | 1.37 (0.20) | 1.19 (0.30)
  BDNF | 37.78 (6.72) | 34.00 (7.44)
  GSK-3b | 20.89 (7.88) | 19.49 (6.47)
  XBP1 | 1.11 (0.36) | 0.96 (0.20)
  MARCKS | 1.32 (0.35) | 1.28 (0.54)
  p-GSK 3b | 4.01 (0.78) | 4.11 (1.54)
  p-GSK 3ab | 2.29 (0.64) | 1.93 (0.55)
  Fyn | 33.01 (5.42) | 30.24 (6.44)
  Timeless | 1.41 (0.12) | 1.42 (0.40)
  PGM1 | 30.96 (4.57) | 28.58 (6.64)
  NFKB p-P65 | 15.03 (6.01) | 14.58 (8.01)
  Calmodulin | 34.44 (5.68) | 31.86 (7.70)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Lithium
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 20/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lithium (N=24)
Increased Thirst (General disorders) | 6
Dry Mouth (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Cognitive Impairment (Psychiatric disorders) | 1
Stomach Upset (Gastrointestinal disorders) | 1
Increased Daytime Sleepiness (General disorders) | 1
Blurred Vision (Eye disorders) | 1
Dizziness (General disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Decreased Sexual Interest (Reproductive system and breast disorders) | 1
Hair Loss (General disorders) | 1
Increased urination (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT02909504/Prot_SAP_000.pdf